CLINICAL TRIAL: NCT00396682
Title: Elimination of CD4+CD25+ Regulatory T Cells in Patients With Advanced HCC After Treatment With Cyclophosphamide
Brief Title: Elimination of CD4+CD25+ Regulatory T Cells in Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Tim Greten, Med. Hochschule Hannover
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAN-HCC-002; DFG - KFO 119
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Advanced HCC
Keywords: HCC; T cell
MeSH Terms: interventions — Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — 150 - 250 - 350 mg

SUMMARY:
It has been shown that patients with advanced HCC have an increased frequency of CD4+CD25+ regulatory T cells. These cells might suppress tumor-specific immune responses. Cyclophosphamide has been shown to reduce the frequency of CD4+CD25+ regulatory T cells. The aim of this study is to test if the treatment with cyclophosphamide leads to a decrease in the frequency of CD4+CD25+ regulatory T cells and to increase tumor specific immune responses in patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* adequate WBC
* adequate liver and kidney function
* no immunodeficiency
* ECOG < 2

Exclusion Criteria:

* advanced liver cirrhosis
* severe cardiopulmonary diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Frequency of CD4+CD25+regulatory T cells | within 8 weeks
Tumor specific immune responses | within 12 weeks

SECONDARY OUTCOMES:
Toxicity | within 8 weeks
Function and Phenotype of CD4+CD25+ regulatory T cells | within 12 weeks
Tumor response | within 12 weeks
Survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — Department of Gastroenterology, Medizinische Hochschule Hannover; Tim F Greten, M.D., Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Germany

REFERENCES:
- [Derived] Greten TF, Ormandy LA, Fikuart A, Hochst B, Henschen S, Horning M, Manns MP, Korangy F. Low-dose cyclophosphamide treatment impairs regulatory T cells and unmasks AFP-specific CD4+ T-cell responses in patients with advanced HCC. J Immunother. 2010 Feb-Mar;33(2):211-8. doi: 10.1097/CJI.0b013e3181bb499f. PMID 20139774